CLINICAL TRIAL: NCT01179100
Title: The Effects Of Lidocaine Infusion On The Recovery Of Cognitive Function Following General Anesthesia In Elderly Patients Undergoing Orthopedic Surgeries Requiring A Minimum Two Day Hospitalization
Brief Title: How Lidocaine Affects Outcomes In Orthopedic Surgery Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Patient population require high amount of opioids.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: Pro00019834
Record Dates: First submitted 2010-04-23; First posted 2010-08-11 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: General Anesthesia; Surgeries Requiring A Minimum One Day Hospitalization; Elderly
Keywords: elderly; general anesthesia; lidocaine infusion; lidocaine; local anesthetic; pain management; cognitive function
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): Normal Saline: Calculated and adjusted to match loading dose and infusion rate of lidocaine equivalent adjusted for weight.
  Interventions: Drug: Lidocaine
- Lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine (10mg/ml) Loading: 1.5 mg/kg + Infusion: 0.035 mg/kg/min

SUMMARY:
This study will evaluate the effect of intraoperative lidocaine infusion on postoperative orientation and concentration in elderly patients having general anesthesia for orthopedic surgeries requiring a minimum 2 days hospitalization.

This study will also aim to determine whether intraoperative lidocaine infusion during general anesthesia improves recovery and patient outcome, as well as to determine whether lidocaine infusion decreases postoperative opioid (pain medication) usage.

DETAILED DESCRIPTION:
Advances in surgical techniques and anesthetic care have resulted in a substantial reduction in peri-operative morbidity and mortality in the elderly. However, post-operative cognitive dysfunction (POCD), as well as episodic post-operative delirium, are still recognized as significant complications following surgery in the elderly. Post-operative cognitive dysfunction is characterized by impairment of memory, concentration, language, comprehension, and social integration. Conversely, post-operative delirium is characterized by intermittent, short-term impaired cognition, disorientation, and abnormalities in memory and perception, which has been shown to lead to increased morbidity and mortality, delayed functional recovery, and prolonged hospital stays. Elderly patients are particularly sensitive to the central nervous system effects of many peri-anesthetic drugs, including benzodiazepines, barbiturates, opioids, and volatile anesthetics, which may play a role in POCD and consequent patient outcomes. Randomized clinical trials have demonstrated no difference in the recovery of cognitive function between commonly used volatile anesthetic agents.

Several simple, bedside tests are available to assess cognitive function and differentiate between cognitive dysfunction and an episode of delirium. The Confusion Assessment Method (CAM) is a standardized rating of delirium that has been validated and has high inter-observer reliability. The CAM criteria are the most commonly used method for diagnosing delirium in hospitalized patients. The Mini-Mental Status Examination (MMSE) and the Abbreviated Mental Test are tools used to assess cognitive function at the bedside.

Lidocaine is one of the most commonly used sodium-channel blockers in the medical armamentarium. It has long been used for its local anesthetic and anti-arrhythmic properties, and has been studied as an adjunct to general anesthesia. While lidocaine is cardio-toxic in excessive doses, the therapeutic and toxic levels are well-documented and wide, making lidocaine a drug with a favorable safety profile. Randomized clinical trials have shown perioperative lidocaine infusions to decrease postoperative pain scores, reduce postoperative opioid requirements, shortens hospital stays, improves postoperative recovery and fatigue score when administered as an adjuvant during surgery. Lidocaine has analgesic, antihypertensive, and anti-inflammatory properties. To date, no clinical trials have been conducted to establish the relationship between lidocaine infusions and postoperative recovery, particularly cognitive function, in elderly orthopedic surgery patients. It is therefore the aim of this study to evaluate the effects of lidocaine infusion on postoperative cognitive function in elderly patients having general anesthesia for orthopedic surgery, and to assess whether intraoperative lidocaine infusion decreases postoperative opioid usage and improves recovery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo orthopedic surgery under general anesthesia requiring a minimum two-day hospitalization (e.g. THA, TKA, hardware removal)
* 65 years of age or older
* ASA Physical Classification I - IV
* Willingness and ability to sign an informed consent document
* English-speaking

Exclusion Criteria:

* Inability to consent or complete cognitive assessments
* Inability to use a PCA system
* Allergy to lidocaine or any other medication administered as part of this protocol
* Emergency surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Post-operative cognitive function | 1 month
  Pre-operative cognitive function tests, including the CAM, MMSE, and the Abbreviated Mental Test, will be administered to establish baseline cognitive function. Then compared with the results of the postoperative cognitive function tests.

SECONDARY OUTCOMES:
Postoperative pain | 1 month
  The postoperative pain will be measured during one month, using follow up questionnaires at 1, 2, or 3, then 7and 30 days after surgery
Opioid consumption obtained from the recorded data | 1 month
  Perioperative use of opioid consumption inside hospital (recorded by study staff and data obtained from patient charts) Post discharge use of opioid consumption (data obtained from the follow up questionnaires at 1, 2, or 3, then 7 and 30 days after surgery)
Postoperative nausea and vomiting using a Verbal Rating Scale | 1 month
  Nausea and vomiting will be measured with follow up questionnaires at 1, 2, or 3, then 7 and 30 days after surgery
Return to normal activities of daily living using follow up questionnaires Return to normal activities of daily living using follow up questionnaires | 1 month
  Return to normal activities of daily living(including dietary intake, bowel and bladder function, physical activities)will be measured in both groups.
Patient satisfaction using a verbal rating scale from 0 to 100 | 1 month
  0= Not satisfied 100= Excellent
Hospital stay | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States